CLINICAL TRIAL: NCT01545492
Title: CHIPS-Child:Testing the Developmental Origins Hypothesis
Brief Title: Testing the Developmental Origins Hypothesis
Acronym: CHIPS-Child
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Laura Magee, Clinical Professor of Medicine, Children's & Women's Health Centre of British Columbia
Other Study IDs: H08-00882CHIPS-Child
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes; Stroke; Obesity
Keywords: CHIPS; famine; reprogramming; developmental; blood; pressure; randomised; randomized; hypertension; anthropometry; measurement; genetics; epigenetics; methylation; cortisol; stress; DNA; growth; weight; length; height
MeSH Terms: conditions — Diabetes Mellitus; Stroke; Obesity; Hypertension; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. ~150 strands of hair
  2. Four buccal swabs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tight: Children born to women in the CHIPS RCT randomized to "Tight" blood pressure control [target diastolic BP 85mmHg]
- Less Tight: Children born to women in the CHIPS RCT randomized to "Less Tight" [target diastolic BP 100mmHg].

SUMMARY:
INTRODUCTION: CHIPS-Child is a parallel, ancillary study to the CHIPS randomized controlled trial (RCT). CHIPS is designed to determine whether 'less tight' control [target diastolic BP (dBP) 100mmHg] or 'tight' control [target dBP 85mmHg] of non-proteinuric hypertension in pregnancy is better for the baby without increasing maternal risk.

CHIPS-Child is a follow up study at 12 m corrected post-gestational age (± 2 m) limited to non-invasive examination [anthropometry, hair cortisol, buccal swabs for epigenetic testing and a maternal questionnaire about infant feeding practices and background]. Annual contact will be maintained in years 2-5 and contact will include annual parental measurement of the child's height, weight and waist circumference.

OBJECTIVE: To directly test, for the first time in humans, whether differential blood pressure (BP) control in pregnancy has developmental programming effects, independent of birthweight. We predict that, like famine or protein malnutrition, 'tight' (vs. 'less tight') control of maternal BP will be associated with fetal under-nutrition and effects will be consistent with developmental programming.

DETAILED DESCRIPTION:
INTRODUCTION: Growing evidence shows that reduced fetal growth rate is associated with adult cardiovascular risk markers (e.g., obesity) and disease, and evidence worldwide indicates that this relationship is independent of birthweight. The leading theory describes 'developmental programming' in utero leading to permanent alteration of the fetal genome. While those changes are adaptive in utero, they may be maladaptive postnatally.

OBJECTIVE: To directly test, for the first time in humans, whether differential blood pressure (BP) control in pregnancy has developmental programming effects, independent of birthweight. We predict that, like famine or protein malnutrition, 'tight' (vs. 'less tight') control of maternal BP will be associated with fetal under-nutrition and effects will be consistent with developmental programming.

METHODS: CHIPS-Child is a parallel, ancillary study to the CHIPS randomized controlled trial (RCT). CHIPS is designed to determine whether 'less tight' control [target diastolic BP (dBP) 100mmHg] or 'tight' control [target dBP 85mmHg] of non-proteinuric hypertension in pregnancy is better for the baby without increasing maternal risk.

CHIPS-Child is a follow up study at 12 m corrected post-gestational age (± 2 m) limited to non-invasive examination [anthropometry, hair cortisol, buccal swabs for epigenetic testing and a maternal questionnaire about infant feeding practices and background]. Annual contact will be maintained in years 2-5 and contact will include annual parental measurement of the child's height, weight and waist circumference.

Sample size:. CHIPS will recruit 1028 women. We estimate that 80% of CHIPS centres will participate in CHIPS-Child, approximately 97% of babies will survive, and 90% of children will be followed to 12 m resulting in a sample size of 626. Power will be >80% to detect a between-group difference of ≥0.25 in 'change in z-score for weight' between birth and 12 m (2-sided alpha=0.05, SD 1).

ELIGIBILITY:
Inclusion Criteria:

* All women participating in CHIPS and their children born after recruitment.

Exclusion Criteria:

* Women who have experienced the loss of their pregnancy or child after recruitment into CHIPS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only women participating in the CHIPS RCT and their children born after recruitment are eligible to participate in CHIPS-Child.
Sampling Method: Non-Probability Sample
Enrollment: 626 (Estimated)
Dates: Start 2012-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
difference in 'change in z score for weight' at 12 m(+/- 2m) | birth to 12m (+/-2m) of age, 24m, 36m, 48m, 60m
  Between-group difference in early postnatal weight gain ('change in z score for weight') between birth and 12 m (p<0.05), 24m, 36m, 48m & 60m.

SECONDARY OUTCOMES:
hypothalamic pituitary adrenal axis function | average of 12m (+/-2m) of age
  Hair collected at 12m (+/-2m) of age will be analysed for hypothalamic pituitary adrenal axis function (hair cortisol for overall cortisol production).
differences in DNA methylation | average of 12 m (+/- 2m) of age
  Buccal swab samples collected at 12m (+/-2m) of age will be assessed for between-groups differences in DNA methylation, using targeted (genes associated with growth, obesity, cardiovascular disease, and/or a developmental programming effect) and global (genome-wide microarray) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Magee, MD, Principal Investigator — BC Children & Women's Health Centre
Locations (41):
- United States (4):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Norton Hospital Downtown & Suburban, Louisville, Kentucky
  - Copper University Hospital, Camden, New Jersey
  - Oregon Health & Science University, Portland, Oregon
- Australia (2):
  - Ipswich Hospital, Ipswich
  - King Edward Memorial Hospital, Subiaco
- Canada (9):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Surrey Memorial Hospital: Jim Pttison Outpatient Care & Surgery Centre, Surrey, British Columbia
  - BC Children & Women's Health Centre, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - CHUS Fleurimont, Sherbrooke, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hopital Sainte-Justine, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Chile (2):
  - Hospital Base Osorno, Osorno
  - Hospital Dr Sotero del Rio, Puente Alto
- Tartu University Hospital - Women's Clinic, Tartu, Estonia
- Netherlands (11):
  - Academic Medical Center, Amsterdam
  - OLVG, Amsterdam
  - VU Medical Center, Amsterdam
  - UMCG, Groningen
  - Tergooiziekenhuizen, Hilversum
  - MUMC Maastricht, Maastricht
  - St Antonius Ziekenhuis, Nieuwegein
  - Diakonessen Ziekenhuis, Utrecht
  - UMCU, Utrecht
  - Maxima Medical Centre, Veldhoven
  - Isala Klinieken Zwolle, Zwolle
- Christchurch Women's Hospital, Christchurch, New Zealand
- United Kingdom (11):
  - Birmingham Women's Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Royal Lancaster Infirmary, Lancaster
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Southport & Ormskirk Hospital, Ormskirk
  - Derriford Hospital, Plymouth
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Singleton Hospital, Swansea
  - New Cross Hospital, Wolverhampton
  - York District Hospital, York

REFERENCES:
- [Background] Wadhwa PD, Buss C, Entringer S, Swanson JM. Developmental origins of health and disease: brief history of the approach and current focus on epigenetic mechanisms. Semin Reprod Med. 2009 Sep;27(5):358-68. doi: 10.1055/s-0029-1237424. Epub 2009 Aug 26. PMID 19711246
- [Background] Waterland RA, Michels KB. Epigenetic epidemiology of the developmental origins hypothesis. Annu Rev Nutr. 2007;27:363-88. doi: 10.1146/annurev.nutr.27.061406.093705. PMID 17465856
- [Background] Gilbert EF, Varakis J, Opitz JM, ZuRhein GM, Ware R, Viseskul C, Kaveggia EG, Hartmann HA. Generalized gangliosidosis type II (juvenile GM1 gangliosidosis). A pathological, histochemical and ultrastructural study. Z Kinderheilkd. 1975 Sep 11;120(3):151-80. doi: 10.1007/BF00439006. PMID 126533
- [Background] Painter RC, Roseboom TJ, Bleker OP. Prenatal exposure to the Dutch famine and disease in later life: an overview. Reprod Toxicol. 2005 Sep-Oct;20(3):345-52. doi: 10.1016/j.reprotox.2005.04.005. PMID 15893910
- [Background] Tobi EW, Lumey LH, Talens RP, Kremer D, Putter H, Stein AD, Slagboom PE, Heijmans BT. DNA methylation differences after exposure to prenatal famine are common and timing- and sex-specific. Hum Mol Genet. 2009 Nov 1;18(21):4046-53. doi: 10.1093/hmg/ddp353. Epub 2009 Aug 4. PMID 19656776
- [Background] Silveira PP, Portella AK, Goldani MZ, Barbieri MA. Developmental origins of health and disease (DOHaD). J Pediatr (Rio J). 2007 Nov-Dec;83(6):494-504. doi: 10.2223/JPED.1728. PMID 18074050
- [Background] Cameron N, Demerath EW. Critical periods in human growth and their relationship to diseases of aging. Am J Phys Anthropol. 2002;Suppl 35:159-84. doi: 10.1002/ajpa.10183. PMID 12653312